CLINICAL TRIAL: NCT07151300
Title: Phonophoresis With Bee Venom: Evaluating Its Efficacy in Managing Pain and Enhancing Mobility in Knee Osteoarthritis Patients
Acronym: BEE-KNEE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU.REC.2025(49H)
Record Dates: First submitted 2025-08-11; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Osteoarthritis
Keywords: Osteoarthritis; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bee Venom Phonophoresis (Experimental): Participants receive bee venom phonophoresis therapy applied to the affected knee(s) using standardized ultrasound parameters. Bee venom topical preparation will be mixed with ultrasound coupling gel and applied to the treatment area. Ultrasound will be delivered at a standardized frequency, intensity, and duration determined before study commencement.
  Interventions: Device: Ultrasound therapy unit; Biological: Bee venom topical preparation (for phonophoresis)
- Control - Placebo Phonophoresis (Placebo Comparator): Participants receive placebo phonophoresis using the same ultrasound parameters as the experimental group, but with a neutral coupling gel that does not contain bee venom. This ensures the same patient experience without the active bee venom component.
  Interventions: Device: Ultrasound therapy unit

INTERVENTIONS:
Device: Ultrasound therapy unit — Ultrasound therapy unit
Biological: Bee venom topical preparation (for phonophoresis) — Bee venom topical preparation (for phonophoresis)
  Arms: Bee Venom Phonophoresis

SUMMARY:
Brief Summary:

This single-blind, randomized controlled trial will investigate the efficacy of bee venom phonophoresis in managing pain and improving mobility in patients with knee osteoarthritis. Thirty adults aged 40-75 years with clinically and radiographically confirmed knee osteoarthritis will be randomly assigned to receive either bee venom phonophoresis or placebo phonophoresis with a neutral gel. Ultrasound parameters will be standardized for all participants.

Primary outcomes are pain reduction, measured by the Visual Analog Scale (VAS), and functional mobility, assessed by the Timed Up and Go (TUG) test. The secondary outcome is walking endurance, measured by the Six-Minute Walk Test (6MWT). Assessments will be conducted at baseline and post-intervention.

The study is designed to determine whether bee venom phonophoresis offers greater clinical benefit compared to placebo phonophoresis, potentially providing a non-invasive, adjunctive treatment option for knee osteoarthritis. Ethical approval has been obtained from the Faculty of Physical Therapy, Sinai University, and all participants will provide written informed consent.

DETAILED DESCRIPTION:
Detailed Description:

Knee osteoarthritis (OA) is a chronic, degenerative joint disease characterized by cartilage loss, joint space narrowing, pain, stiffness, and functional impairment. It is a leading cause of disability worldwide, particularly among older adults. Conventional management includes pharmacologic interventions such as oral analgesics and nonsteroidal anti-inflammatory drugs, and non-pharmacologic approaches such as exercise therapy and physiotherapy. However, these treatments may not provide adequate symptom relief and can be associated with side effects, prompting the search for alternative or adjunctive therapies.

Phonophoresis, an ultrasound-based technique that enhances transdermal drug delivery, has been investigated as a non-invasive intervention for musculoskeletal pain management. Bee venom, used in traditional medicine for inflammatory and arthritic conditions, possesses anti-inflammatory, analgesic, and immunomodulatory properties. Combining bee venom with phonophoresis may enhance penetration into periarticular tissues, potentially improving clinical outcomes in OA patients.

This single-blind, randomized controlled trial will enroll 30 adults aged 40-75 years with clinically and radiographically confirmed knee osteoarthritis. Participants will be randomly allocated to one of two groups:

Experimental group: Bee venom phonophoresis using standardized ultrasound parameters (frequency, intensity, duration).

Control group: Placebo phonophoresis using identical ultrasound settings but with a neutral gel lacking bee venom.

Primary outcomes include pain reduction assessed by the Visual Analog Scale (VAS) and functional mobility assessed by the Timed Up and Go (TUG) test. The secondary outcome is walking endurance, measured by the Six-Minute Walk Test (6MWT). Outcomes will be evaluated at baseline and after the intervention period.

Data will be analyzed using appropriate descriptive and inferential statistics, with between-group comparisons conducted using independent t-tests or nonparametric equivalents, and within-group comparisons using paired t-tests or Wilcoxon signed-rank tests. Statistical significance will be set at p < 0.05.

Ethical approval has been obtained from the Faculty of Physical Therapy, Sinai University. Written informed consent will be obtained from all participants before enrollment. The trial will adhere to the principles of the Declaration of Helsinki and ICH-GCP guidelines to ensure participant safety, data integrity, and scientific validity.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Clinically and radiographically confirmed knee osteoarthritis
* Moderate to severe pain (VAS ≥ 4)
* Willingness to provide informed consent

Exclusion Criteria:

* Allergy to bee products or topical agents used in the study
* Knee surgery or trauma in the past year
* Intra-articular injection in the past 6 months
* Other musculoskeletal or systemic conditions affecting the knees (e.g., rheumatoid arthritis)
* Pregnancy or contraindication to ultrasound therapy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain severity.
Change in Functional Mobility | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using the Timed Up and Go (TUG) test, which records the time (in seconds) taken for a participant to stand up from a chair, walk 3 meters, turn, return, and sit down. Lower times indicate better mobility.

SECONDARY OUTCOMES:
Change in Walking Endurance | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using the Six-Minute Walk Test (6MWT), recording the total distance (in meters) walked in six minutes on a flat surface. Greater distances indicate improved endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai university, Cairo, Egypt